CLINICAL TRIAL: NCT02879877
Title: A Subject-blind, Investigator-blind, Randomized, Placebo-controlled, First-in-human Study Evaluating the Safety/Tolerability, Pharmacokinetics, Effect on Transglutaminase 2 Expression, and Occupancy of Single Ascending Intravenous and Subcutaneous Doses of UCB7858 in Healthy Subjects
Brief Title: A First-In-Human Study With a Single Ascending Dose of UCB7858 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0029; 2016-001129-15 (EudraCT Number)
Record Dates: First submitted 2016-07-29; First posted 2016-08-26 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Healthy Volunteers
Keywords: First in human; subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- UCB7858 (intravenous) (Experimental): Various single doses, administered to various cohorts.
  Interventions: Drug: UCB7858
- Placebo (intravenous) (Placebo Comparator): Single dose placebo comparator for each cohort of iv administration.
  Interventions: Drug: Placebo
- UCB7858 (subcutaneous) (Experimental): Various single doses, administered to various cohorts.
  Interventions: Drug: UCB7858
- Placebo (subcutaneous) (Placebo Comparator): Single dose placebo comparator for each cohort of sc administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UCB7858
  Arms: UCB7858 (intravenous); UCB7858 (subcutaneous)
Drug: Placebo
  Arms: Placebo (intravenous); Placebo (subcutaneous)

SUMMARY:
This study is designed to evaluate the safety and tolerability of UCB7858 when given as single ascending doses administered by intravenous or subcutaneous infusion in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers who gave their written consent by signing the Informed Consent Form
* Subjects in the age between 18 and 55 years old with normal weight as determined by a body mass index (BMI) between 18 and 30 kg/m^2, with a body weight of at least 50 kg for male subjects or 45 kg for female subjects
* Subject has clinical laboratory test results within the reference ranges of the testing laboratory or outside the reference range of the laboratory but considered as not clinically significant by the Investigator
* Subjects has blood pressure (BP) and pulse within normal range in a supine position after 5 minutes rest
* Subject's electrocardiogram (ECG) is considered normal or abnormal but clinically non significant
* Female subjects of childbearing potential must agree to use a highly effective method of birth control during the study and for a period of 6 months after dosing of IMP

Exclusion Criteria:

* Subject has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the subject's ability to participate in this study: Subject has any acute or chronic illness which, in the opinion of the Investigator, may place the subject at risk because of participation in the study. Subject has any clinically relevant abnormal findings in physical examination, laboratory tests, vital signs, or ECG, which, in the opinion of the Investigator, may place the subject at risk because of participation in the study.
* Tests positive for Human Immunodeficiency Virus (HIV)-1 or-2 antibodies, Hepatitis B Virus (HBV) surface antigen, or Hepatitis C Virus (HCV) antibody at Screening
* Any of the following hematological function tests at the Screening Visit: Hemoglobin <111g/L (for women) or <113g/L (for men)
* Absolute neutrophil count <1.5x10^9/L (<1000/mm^3); Platelets <150x10^9/L
* Female subject who is breastfeeding, pregnant, or plans to become pregnant during the study or within 6 months following the final dose of the IMP

For subjects enrolled in the cohorts where the skin biopsies will be performed (Cohort 7 onward), the following exclusion criteria will also apply:

* Subject has a known hypersensitivity to dressings, local anesthetics, suture material, or relevant local/oral antibiotic therapy
* Subject has or had a history of a known inflammatory dermatological condition including eczema, atopic dermatitis, candidiasis, psoriasis, recurrent or persistent fungal infection, or bacterial infections
* Subject uses steroid or nonsteroidal anti-inflammatory drug (NSAID)-containing skin creams on a regular basis
* Subject has used NSAID or NSAID-containing medications within 7 days of randomization
* Subject has used skin emollients within 7 days of randomization on the area of the skin from buttocks
* Subject has tattoos, nevi, or other skin abnormalities such as keloids (or history of keloids, folliculitis, or acne vulgaris) that may, in the opinion of the Investigator, interfere with study assessments.
* Subject has been participating in recreational sun-bathing, or use of sun-bed, on the area of the skin from buttocks within 7 days of Screening
* Subject has active neoplastic disease or history of neoplastic disease within 5 years of the Screening Visit
* Subject has a history of moderate to severe allergic reaction to medication(s) including biologics (for subjects in Cohort 11 only).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events following administration of UCB7858 | Cohort 1-10: Day 1 up to Day 72 Cohort 11: Day 1 up to Day 120

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Cohort 1-10: Predose (Day 1) up to Day 72 Cohort 11: Predose (Day 1) up to Day 120
Time to reach Cmax (tmax) | Cohort 1-10: Predose (Day 1) up to Day 72 Cohort 11: Predose (Day 1) up to Day 120
Area under the curve from time 0 to time t, the time of last quantifiable concentration [AUC(0-t)] | Cohort 1-10: Predose (Day 1) up to Day 72 Cohort 11: Predose (Day 1) up to Day 120
Area under the curve from 0 to infinity (AUC) | Cohort 1-10: Predose (Day 1) up to Day 72 Cohort 11: Predose (Day 1) up to Day 120
The terminal plasma half-life (t1/2) following intravenous administration | Cohort 1-10: Predose (Day 1) up to Day 72 Cohort 11: Predose (Day 1) up to Day 120
Plasma clearance (CL) of UCB7858 following intravenous administration | Cohort 1-10: Predose (Day 1) up to Day 72 Cohort 11: Predose (Day 1) up to Day 120
Volume of distribution (Vss) for UCB7858 at steady state following intravenous administration | Cohort 1-10: Predose (Day 1) up to Day 72 Cohort 11: Predose (Day 1) up to Day 120
Apparent volume of distribution (Vss/F) of UCB7858 following subcutaneous administration | Cohort 1-10: Predose (Day 1) up to Day 72 Cohort 11: Predose (Day 1) up to Day 120
Apparent plasma clearance (CL/F) of UCB7858 following subcutaneous administration | Cohort 1-10: Predose (Day 1) up to Day 72 Cohort 11: Predose (Day 1) up to Day 120
Mean absolute bioavailability (F) of UCB7858 given subcutaneously, using the ratio of geometric mean AUCs for subcutaneous (sc) administration and intravenous (iv) infusion (AUC_sc/AUC_iv) | Cohort 1-10: Predose (Day 1) up to Day 72 Cohort 11: Predose (Day 1) up to Day 120
Concentration of UCB7858 at the end of infusion (Cinf) | Cohort 1-10: Predose (Day 1) up to Day 72 Cohort 11: Predose (Day 1) up to Day 120
Time at the end of infusion of UCB7858 (tinf) | Cohort 1-10: Predose (Day 1) up to Day 72 Cohort 11: Predose (Day 1) up to Day 120

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (+1 844 599 2273)
Locations (1):
- Up0029 001, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, Individual Patient Data cannot be adequately anonymized and there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.